CLINICAL TRIAL: NCT01480492
Title: Study the Effect of Nucleoside on Host Immune in Patients With CHB
Brief Title: Effect of Antiviral Therapy on Host Immune in Patients With Chronic Hepatitis B Virus(HBV) Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cz Li (Other)
Responsible Party: Sponsor-Investigator, Cz Li, professor, Changhai Hospital
Organization: Changhai Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HBV20111115; 09zr400500 (Other Grant/Funding Number: Shanghai Natural Science Fund); 30972600 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2011-11-15; First posted 2011-11-29 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: HBeAg Positive Chronic Hepatitis B Infection
Keywords: HBV; Immune; antiviral therapy
MeSH Terms: interventions — Telbivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- therapy (No Intervention)
  Interventions: Drug: Telbivudine

INTERVENTIONS:
Drug: Telbivudine — 600mg,1/d,one year

SUMMARY:
During hepatitis B virus(HBV) infection host immune plays important role.Recently there are many different antiviral therapy methods.Different antiviral therapy methods showed different effector.In order to investigate whether these antiviral therapy methods especially methods directly inhibit viral replication have some effect on host immune the investigators designed these study. The investigators want to observe the change of host immune during antiviral therapy in patients with chronic HBV infection, and analyze the relationship between these changes and the antiviral effector of these drugs.

ELIGIBILITY:
inclusion criteria:

* 18-65 years old
* chronic HBV infection
* HBeAg positive,HBV DNA more than 10E5 IU/mL
* ALT ≥2×UTL

exclusion criteria:

* with liver cancer
* with liver failure
* pregnant

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
change of programmed death-1(PD-1) level of patients with chronic HBV infection during therapy | base line-4 weeks-12 weeks-24 weeks-end of therapy

SECONDARY OUTCOMES:
Decline of hepatitis B e antigen (HBeAg) level | base line-4weeks-12weeks-24weeks-end of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Wan Mo Bin, Professor, Study Director — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Li CZ, Hu JJ, Xue JY, Yin W, Liu YY, Fan WH, Xu H, Liang XS. Viral infection parameters not nucleoside analogue itself correlates with host immunity in nucleoside analogue therapy for chronic hepatitis B. World J Gastroenterol. 2014 Jul 28;20(28):9486-96. doi: 10.3748/wjg.v20.i28.9486. PMID 25071343